CLINICAL TRIAL: NCT00945464
Title: Scripps Polster Breast Care Center Investigational GeneBank
Acronym: PINK
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: LAJ 08-8001
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Approximately 19.5 mls of blood will be collected from volunteers. The blood from each subject will be collected via venipuncture. If subject is unable/unwilling to provide blood sample, we can also collect 2 mls of saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Women over the age of 30 undergoing breast imaging at the Scripps Polster Breast Care Center.
  Interventions: Other: Blood/saliva samples, historic breast imaging

INTERVENTIONS:
Other: Blood/saliva samples, historic breast imaging — Subjects are required only to provide a blood or saliva sample, relevant personal and family history (if available), and 5 years of historic breast imaging reports.

SUMMARY:
Breast cancer is a disease of complex origin with a strong genetic component. The incidence of breast cancer is very high in monozygotic twins of patients, and it is thought that a high proportion and perhaps the majority of breast cancers arise in a small number of genetically susceptible women. Recent studies in human genetics have discovered several intervals in the human genome containing inherited variants that are statistically associated with the propensity to develop breast cancer. The investigators plan to use this knowledge to design a genetic screening test to guide recommendations for breast cancer screening with mammography. If the small group of genetically susceptible women can be identified, more effective breast cancer screening strategies can be implemented. In contrast, a very large proportion of women who undergo yearly mammography are at exceptionally low risk from a genetic perspective. Using genomic guidance could eventually reconfigure the most efficacious strategy to screen women for early detection of breast cancer.

By developing a genetic screening panel based on genetic markers for breast cancer, the investigators will be able to more accurately determine a woman's individual risk for developing breast cancer.

DETAILED DESCRIPTION:
Women the age of 30 or over who are undergoing screening or diagnostic breast imaging as an out patient at the Scripps Polster Breast Care Center in La Jolla, CA, with at least 5 years of historic breast imaging data available will be eligible to enroll. For this study, consecutive subjects who have completed screening or diagnostic breast imaging at the Scripps Polster Breast Care Center will be enrolled for one day. It is estimated that up to 5000 subjects will be included in the cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 years or older
2. Be reliable, cooperative and willing to comply with all protocol-specified procedures
3. Able to understand and grant informed consent
4. Be undergoing screening or diagnostic breast imaging
5. Have at least 5 years of breast imaging data available

Exclusion Criteria:

1. Have a significant chronic medical condition which, in the Investigator's opinion, would interfere with the subject's participation in the study
2. Have undergone treatment with any investigational agents or devices within thirty days preceding enrollment in the study
3. Have taken any CNS sedation or depressants in past 12 hours

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women over the age of 30 undergoing breast imaging at the Scripps Polster Breast Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 1136 (Actual)
Dates: Start 2008-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Genotyping | End of study
  Genotype a panel of single nucleotide polymorphisms (SNPs) previously shown to be highly associated with increased risk to breast cancer in a cohort of women with either at least 5 years of historical breast imaging data available or 30-45 year old breast cancer patients with at least one year imaging data

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Topol, MD, Principal Investigator — Scripps Translational Science Institute and Genomic Medicine
Locations (1):
- Scripps Polster Breast Care Center, La Jolla, California, United States